CLINICAL TRIAL: NCT01580046
Title: Renal Toxicity of Iodixanol and Iopromide in Patients With Renal Dysfunction-a Multicentre, Single Blind, Randomized Controlled, Prospective Trial
Brief Title: Renal Toxicity of Iodixanol and Iopromide in Patients With Renal Dysfunction
Acronym: RIPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Huo (Other)
Responsible Party: Sponsor-Investigator, Yong Huo, MD, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XNK201201
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Kidney Failure, Chronic
Keywords: Chronic Kidney Disease; Coronary Angiography; Contrast Media; Percutaneous Coronary Intervention; Serum Creatinine; Glomerular Filtration Rate; Iodixanol; Iopromide
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — iodixanol; iopromide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iodixanol (Experimental)
  Interventions: Drug: iodixanol
- iopromide (Active Comparator)
  Interventions: Drug: iopromide

INTERVENTIONS:
Drug: iodixanol — 1. coronary angiography, 32gI/100ml, 40～60 ml once injection
  2. left ventricular, aortic root and selective coronary angiography, 32gI/100ml, 30～60 ml once injection
  Arms: Iodixanol
Drug: iopromide — coronary angiography, 370mgI/ml(0.769gIopromide/ml),5～8 ml once injection
  Other Names: Ultravist
  Arms: iopromide

SUMMARY:
The purpose of this study is to compare renal toxicity of Iodixanol and Iopromide in patients with renal dysfunction.

DETAILED DESCRIPTION:
The study is designed to compare renal toxicity of Iodixanol and Iopromide after coronary angiography or percutaneous coronary intervention (PCI) in patient with Chronic Kidney Disease, considering original renal function and adequate hydration. The risk of varying degree of renal impairment, changes of serum Cys C level will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Provides written Informed Consent and is willing to comply with protocol requirements
* Is referred for cardiac angiography, with or without PCI
* Has a documented predose serum creatinine level of 1.5～3.5 mg/dl for men and 1.3～3.0 mg/dl for women
* Serum creatinine levels of twice tests conform with the baseline criteria, and the difference of twice serum creatinine tests is not more than 30%(first test: within 3 month,prior to enrollment; second test: at enrollment)

Exclusion Criteria:

* Has a history of hypersensitivity to iodine-containing compounds
* Has end-stage renal disease
* Has kidney transplantation
* Has creatinine clearance rates >60 ml/min in last 3 months
* Has acute coronary syndrome with heart failure(above class II in accordance with Killip or class III in accordance with the classification of the New York Heart Association (NYHA)) and shock
* Patients with cancer
* Has diabetes with serious complications, other kidney organs
* Patients with serious blood system disease
* Heart failure [class III~Ⅳ in accordance with the classification of the New York Heart Association (NYHA) and (or) pulmonary edema]
* Patients with hepatic insufficiency[3 times as ALT and (or) AST normal reference value limit]
* Has received an iodinated contrast agent within 14 days prior to the administration of the study agent
* Is scheduled to receive an iodinated contrast agent within 7 days after administration of the study agent
* Has acute renal failure or end-stage renal disease requiring dialysis in the past 3 months
* Use of 3 days continuously nonsteroidal anti-inflammatory drugs within 1 week of the procedure
* Patients with hypotension [(SBP<80 mmHg for over 1h and needing Medication or intraaortic balloon counterpulsation(IABP) ]
* Uncontrolled condition of hyperthyroidism
* pregnancy or lactation
* Is planned to receive the drugs without permission in this protocol
* Participating in another intervention research study in last 3 months
* legally incapacitated or limitations
* Any other conditions not suitable to be enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
to evaluate the change in Glomerular Filtration Rate levels by Estimated Glomerular Filtration Rate | days 3 and 7

SECONDARY OUTCOMES:
In each group(Iodixanol group and Iopromide group), the proportion of patients exhibiting an increases of serum creatinine in different range(<10%,10%~25%, and ≥25%), comparing with baseline level. | days 3 and 7
Incidence of hemodialysis | days 3 and 7
Changes of Cystatin C level from baseline | days 1 and 3

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Academy Of Medical Sciences Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangxi Medical University, Nanning, Guangxi
  - The People's Hospital Of Hebei Province, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Luoyang, Henan
  - The Second Affiliated Hospital To Nanchang University, Nanchang, Jiangxi
  - The People's Hospital Of Liaoning Province, Shenyang, Liaoning
  - The Affiliated Hospital Of Medical College Qingdao University, Qingdao, Shandong
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Peking University People's Hospital, Beijing
  - Pla Navy General Hospital, Beijing
  - The Central Hospital Of China Aerospace Corporation, Beijing
  - Chinese PLA General Hospital, Beijing
  - Xinqiao Hospital, Third Military Medical University, Chongqing
  - Renji Hospital ，Shanghai Jiao Tong University School Of Medicine, Shanghai
  - Shanghai Chest Hospital Affiliated To Shanghai Jiaotong University, Shanghai
  - Shanghai First People's Hospital, Shanghai